CLINICAL TRIAL: NCT02528422
Title: The Effect of Acyl-Ghrelin on Kidney Function and Blood Pressure in Healthy Volunteers - A Randomized, Cross-over, Single-blind, Placebo-controlled Dose-response Study of the Acyl-ghrelin Induced Effects on GFR, Tubular Transport of Sodium and Water in Different Nephron Segments and Central and Peripheral Blood Pressure
Brief Title: The Effect of Acyl-Ghrelin on Kidney Function and Blood Pressure in Healthy Volunteers
Acronym: DOAG
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Erling Bjerregaard Pedersen (Other)
Collaborators: University of Aarhus (Other)
Responsible Party: Sponsor-Investigator, Erling Bjerregaard Pedersen, Professor, MD, Dr.Sci., Regional Hospital Holstebro
Organization: Regional Hospital Holstebro (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: MY-1-2014; 2014-004496-23 (EudraCT Number)
Record Dates: First submitted 2015-08-17; First posted 2015-08-19 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Renal Tubular Transport
MeSH Terms: interventions — acyl-ghrelin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 50 µg Acyl-Ghrelin (Active Comparator): Intravenous injection on examination day.
  Interventions: Drug: Acyl-Ghrelin
- 100 µg Acyl-Ghrelin (Active Comparator): Intravenous injection on examination day.
  Interventions: Drug: Acyl-Ghrelin
- Isotonic Sodium Chloride (Placebo Comparator): Intravenous injection on examination day.
  Interventions: Drug: Acyl-Ghrelin

INTERVENTIONS:
Drug: Acyl-Ghrelin

SUMMARY:
Ghrelin (growth hormone release inducer) is produced in the stomach. The active form of Ghrelin is Acyl-Ghrelin. Acyl-Ghrelin stimulates the Ghrelin receptors. Ghrelin receptors are detected in the distal tubules in mice and animal studies have shown that Ghrelin increases the absorption of sodium in the renal tubules. Ghrelin infusion directly into the renal artery of rats increased sodium reabsorption in the distal nephron, presumably via the epithelial sodium channels (ENaC).

The purpose of the study is to measure the acyl-ghrelin induced effects on GFR, tubular transport of sodium and water in different nephron segments and central and peripheral blood pressure in a randomized, cross-over, single-blind, placebo-controlled dose-response study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40 years,
* BMI 18,5-30kg/m2,
* women must use contraception.

Exclusion Criteria:

* Tobacco smoking,
* substance abuse,
* consumption of more than 7 units of alcohol/week for women and more than 14 units/week for men,
* medical treatment except for contraception,
* pregnancy or nursing,
* allergy to acyl-ghrelin,
* significant clinical signs of heart-, lung-, liver-, kidney-, endocrine-, brain- or neoplastic disorders,
* clinically significant abnormal findings in screening blood samples,
* urine sample or ECG,
* office blood pressure over 140/90 mmHg,
* donation of blood within 1 month of the first day of investigation.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2015-05; Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Fractional sodium excreation (FENa) | 5-6 Hours
  Measurement of FENa at baseline and after Acyl-Ghrelin injection

SECONDARY OUTCOMES:
Renal function | 5-6 Hours
  Measurement of GFR, FEK and CH20 at baseline and after Acyl-Ghrelin injection
Water and sodium transport | 5-6 Hours
  Measurement of u-AQP2, u-NCC , u-NKCC -2 and u-ENaC at baseline and after Acyl-Ghrelin
Vasoactive hormones | 5-6 Hours
  Measurement of p-BNP , PRC, p-AngII , p-Aldo and p-AVP at baseline and after Acyl-Ghrelin
Blood pressure | 5-6 Hours
  Measurement of Central blood pressure, PWV, AIx and Peripheral blood pressure at baseline and after Acyl-Ghrelin

CONTACTS AND LOCATIONS:
Overall Officials: Erling B Pedersen, Study Chair — Department of Medical Research and Medicine, Holstebro Regional Hospital
Locations (1):
- Department of Medical Research, Regional Hospital Holstebro, Holstebro, Denmark